CLINICAL TRIAL: NCT00002602
Title: A PHASE I/II DOSE ESCALATION STUDY USING THREE DIMENSIONAL CONFORMAL RADIATION THERAPY FOR ADENOCARCINOMA OF THE PROSTATE
Brief Title: Radiation Therapy in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9406; CDR0000063854
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Clinical stages T1b-c or T2a-b with PSA + ([Gleason -6] x 10) is ≤ 15. Escalating doses of three dimensional conformal radiation therapy (3D-CRT) until the maximum tolerated dose (MTD) is established.
  Interventions: Radiation: 3D-CRT
- Group 2 (Experimental): Clinical stages T1b-c or T2a-b with PSA + ([Gleason -6]x10)>15. Any clinical T2c with PSA < 70. Must be lymph node negative. Escalating doses of three dimensional conformal radiation therapy (3D-CRT) until the maximum tolerated dose (MTD) is established.
  Interventions: Radiation: 3D-CRT
- Group 3 (Experimental): Clinical stage T3 with PSA < 70. Must be lymph node negative. Escalating doses of three dimensional conformal radiation therapy (3D-CRT) until the maximum tolerated dose (MTD) is established.
  Interventions: Radiation: 3D-CRT

INTERVENTIONS:
Radiation: 3D-CRT — 3 dimensional conformal radiation therapy
  Other Names: 3 dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for prostate cancer.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy in treating patients who have previously untreated stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of 3-dimensional conformal radiotherapy to the prostate gland and immediately surrounding tissues in patients with stage II or III adenocarcinoma of the prostate. II. Determine the normal tissue toxicity rate of this regimen in the rectums and bladders of these patients. III. Determine local control by clinical and pathologic examination and by PSA determinations in patients treated with this regimen. IV. Determine the distant failure and overall survival of patients treated with this regimen.

OUTLINE: This is a dose escalation study. Patients are stratified according to 1 of the following 3 prognostic groups: Group 1: T1b-c or T2a-b with combined PSA/Gleason (CPG) score 15 and under Group 2: T1b-c or T2a-b with CPG score more than 15, or any T2c with PSA less than 70 ng/mL Group 3: T3 with prostate specific antigen (PSA) less than 70 ng/mL Patients receive 3-dimensional (3-D) conformal radiotherapy 5 days a week for 7.6, 8.2, or 8.8 weeks. Cohorts of 120-270 patients receive escalating doses of 3-D conformal radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 20% of patients experience dose-limiting toxicity. Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 549-801 patients (120-204 patients for the first dose level, 237-321 patients for the second dose level, and 192-276 patients for the third dose level) will be accrued for this study within 4.75 to 5.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated adenocarcinoma of the prostate T1b-c or T2a-b with a Gleason score more than 5 and PSA greater than 4 ng/mL OR Any T3 PSA under 70 ng/mL within 3 weeks prior to entry and at least 10 days after prostate biopsy No biopsy proven regional nodal involvement No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Hematopoietic: White blood cell (WBC) count of at least 4,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 11 g/dL Hepatic: Not specified Renal: Not specified Other: No major medical or psychiatric illness that would preclude study No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed Radiotherapy: No prior pelvic irradiation Surgery: No prior prostatectomy or cryosurgery for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Actual)
Dates: Start 1994-05; Primary Completion 2004-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of radiation that can be delivered to the prostate gland and immediate surrounding tissues in patients with carcinoma of the prostate using three dimensional conformal radiation therapy (3D-CRT). | From registration to approximately 18 months from the start of treatment

SECONDARY OUTCOMES:
To quantify the normal tissue toxicity rate (normal tissue complication probability (NTCP)) for rectum and bladder using 3D-CRT | From registration to approximately 18 months from the start of treatment
To evaluate local control by clinical, pathologic, and PSA (stable in normal range) determinations | From registration to the date of progression or last follow-up. Analysis will occur after the primary endpoint analysis.
Distant metastasis and survival | From registration to the date of death or last follow-up. Analysis will occur after the primary endpoint analysis.

CONTACTS AND LOCATIONS:
Overall Officials: James D. Cox, MD, Study Chair — M.D. Anderson Cancer Center
Locations (228):
- United States (213):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Mount Diablo Medical Center, Concord, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Regional Medical Center, Midland, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNIMED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (15):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Du KL, Bae K, Movsas B, Yan Y, Bryan C, Bruner DW. Impact of marital status and race on outcomes of patients enrolled in Radiation Therapy Oncology Group prostate cancer trials. Support Care Cancer. 2012 Jun;20(6):1317-25. doi: 10.1007/s00520-011-1219-4. Epub 2011 Jul 1. PMID 21720747
- [Background] Roach M, Moughan J, Movsas B, et al.: Socio-demographic predictors of biochemical failure and survival among high risk patients treated on Radiation Therapy Oncology Group (RTOG) prostate cancer trials: a meta-analysis. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1127, S204, 2006.
- [Result] Michalski J, Winter K, Roach M, Markoe A, Sandler HM, Ryu J, Parliament M, Purdy JA, Valicenti RK, Cox JD. Clinical outcome of patients treated with 3D conformal radiation therapy (3D-CRT) for prostate cancer on RTOG 9406. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):e363-70. doi: 10.1016/j.ijrobp.2011.12.070. PMID 22633552
- [Result] Tucker SL, Dong L, Michalski JM, Bosch WR, Winter K, Cox JD, Purdy JA, Mohan R. Do intermediate radiation doses contribute to late rectal toxicity? An analysis of data from radiation therapy oncology group protocol 94-06. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):390-5. doi: 10.1016/j.ijrobp.2011.11.073. Epub 2012 Feb 17. PMID 22342302
- [Result] Tucker SL, Michalski JM, Bosch WR, Mohan R, Dong L, Winter K, Purdy JA, Cox JD. Use of fractional dose-volume histograms to model risk of acute rectal toxicity among patients treated on RTOG 94-06. Radiother Oncol. 2012 Jul;104(1):109-13. doi: 10.1016/j.radonc.2012.04.023. Epub 2012 Jun 5. PMID 22673726
- [Result] Tucker SL, Thames HD, Michalski JM, Bosch WR, Mohan R, Winter K, Cox JD, Purdy JA, Dong L. Estimation of alpha/beta for late rectal toxicity based on RTOG 94-06. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):600-5. doi: 10.1016/j.ijrobp.2010.11.080. Epub 2011 Mar 4. PMID 21377288
- [Result] Valicenti RK, Bae K, Michalski J, Sandler H, Shipley W, Lin A, Cox J. Does hormone therapy reduce disease recurrence in prostate cancer patients receiving dose-escalated radiation therapy? An analysis of Radiation Therapy Oncology Group 94-06. Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1323-9. doi: 10.1016/j.ijrobp.2010.01.009. PMID 21414514
- [Result] Michalski JM, Bae K, Roach M, Markoe AM, Sandler HM, Ryu J, Parliament MB, Straube W, Valicenti RK, Cox JD. Long-term toxicity following 3D conformal radiation therapy for prostate cancer from the RTOG 9406 phase I/II dose escalation study. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):14-22. doi: 10.1016/j.ijrobp.2009.01.062. PMID 19577865
- [Result] Tucker SL, Dong L, Bosch WR, Michalski J, Winter K, Mohan R, Purdy JA, Kuban D, Lee AK, Cheung MR, Thames HD, Cox JD. Late rectal toxicity on RTOG 94-06: analysis using a mixture Lyman model. Int J Radiat Oncol Biol Phys. 2010 Nov 15;78(4):1253-60. doi: 10.1016/j.ijrobp.2010.01.069. Epub 2010 Jul 2. PMID 20598811
- [Result] Cheung MR, Tucker SL, Dong L, et al.: Dose-volume analyses of grade ≥ 2 late rectal toxicity among patients treated on protocol RTOG 94-06. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-16, S9, 2007.
- [Result] Tucker SL, Dong L, Bosch WR, et al.: Fit of a generalized Lyman normal-tissue complication probability (NTCP) model to grade ≥ 2 late rectal toxicity data from patients treated on protocol RTOG 94-06. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-15, S8-9, 2007.
- [Result] Valicenti RK, Bae K, Michalski J, et al.: Does adjuvant hormonal therapy improve freedom from biochemical relapse in prostate cancer patients receiving dose- escalated radiation therapy? An analysis of RTOG 94-06. [Abstract] American Society of Clinical Oncology 2007 Prostate Cancer Symposium, 22-24 February 2007, Orlando, FL. A-297, 2007.
- [Result] Michalski JM, Winter K, Purdy JA, Parliament M, Wong H, Perez CA, Roach M, Bosch W, Cox JD. Toxicity after three-dimensional radiotherapy for prostate cancer on RTOG 9406 dose Level V. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):706-13. doi: 10.1016/j.ijrobp.2004.11.028. PMID 15936549
- [Result] Michalski JM, Winter K, Purdy JA, Perez CA, Ryu JK, Parliament MB, Valicenti RK, Roach M 3rd, Sandler HM, Markoe AM, Cox JD. Toxicity after three-dimensional radiotherapy for prostate cancer with RTOG 9406 dose level IV. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):735-42. doi: 10.1016/S0360-3016(03)01578-5. PMID 14967428
- [Result] Roach M, Winter K, Michalski JM, Cox JD, Purdy JA, Bosch W, Lin X, Shipley WS. Penile bulb dose and impotence after three-dimensional conformal radiotherapy for prostate cancer on RTOG 9406: findings from a prospective, multi-institutional, phase I/II dose-escalation study. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1351-6. doi: 10.1016/j.ijrobp.2004.05.026. PMID 15590164
- [Result] Michalski JM, Winter K, Purdy JA, Wilder RB, Perez CA, Roach M, Parliament MB, Pollack A, Markoe AM, Harms W, Sandler HM, Cox JD. Preliminary evaluation of low-grade toxicity with conformal radiation therapy for prostate cancer on RTOG 9406 dose levels I and II. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):192-8. doi: 10.1016/s0360-3016(03)00072-5. PMID 12694838
- [Result] Michalski J, Winter K, Purdy JA, et al.: Toxicity following 3D radiation therapy for prostate cancer on RTOG 9406 dose level V. [Abstract] Int J Radiat Oncol Biol Phys 57 (2 Suppl): S151, 2003.
- [Result] Valicenti RK, Winter K, Cox JD, Sandler HM, Bosch W, Vijayakumar S, Michalski J, Purdy J. RTOG 94-06: is the addition of neoadjuvant hormonal therapy to dose-escalated 3D conformal radiation therapy for prostate cancer associated with treatment toxicity? Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):614-20. doi: 10.1016/s0360-3016(03)00640-0. PMID 14529764
- [Result] Michalski JM, Purdy JA, Winter K, Roach M 3rd, Vijayakumar S, Sandler HM, Markoe AM, Ritter MA, Russell KJ, Sailer S, Harms WB, Perez CA, Wilder RB, Hanks GE, Cox JD. Preliminary report of toxicity following 3D radiation therapy for prostate cancer on 3DOG/RTOG 9406. Int J Radiat Oncol Biol Phys. 2000 Jan 15;46(2):391-402. doi: 10.1016/s0360-3016(99)00443-5. PMID 10661346
- [Result] Roach M, Winter K, Michalski J, et al.: Mean dose of radiation to the bulb of penis correlates with risk of impotence at 24 months: preliminary analysis of Radiation Therapy Oncology Group (RTOG) phase I/II dose escalation trial 94-06. Int J Radiat Oncol Biol Phys 48(3 suppl): A-2104, 316, 2000.
- [Derived] McDonald AM, DeMora L, Yang ES, Hoyle JM, Lenzie A, Williams GR, Michalski JM, Yee D, Bahary JP, Den RB, Roach M 3rd, Dess R, Mishra MV, Valicenti RK, Lau HY, Marcrom SR, Souhami L, Mendez LC, Chen Y, Doncals DE, Pugh SL, Feng FY, Sandler HM. Body composition and mortality in men receiving prostate radiotherapy: A pooled analysis of NRG/RTOG 9406 and NRG/RTOG 0126. Cancer. 2023 Mar 1;129(5):685-696. doi: 10.1002/cncr.34596. Epub 2022 Dec 29. PMID 36579470